CLINICAL TRIAL: NCT06784869
Title: The Efficacy of Scaling and Root Planing on Endothelin-1 Gingival Crevicular Fluid Levels Among Periodontitis Patients: a Randomized Clinical Trial
Brief Title: The Efficacy of Scaling and Root Planing on Endothelin-1 Level
Acronym: clinical
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Sarah Alrihaymee, Head of periodontic department, University of Baghdad
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1/10/2024
Record Dates: First submitted 2025-01-08; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Periodontitis
Keywords: periodontitis; endotheiln-1; scaling and root surface debritment
MeSH Terms: conditions — Periodontitis | interventions — Weights and Measures; Root Planing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- have generalized unstable periodontitis with a moderately deep pocket (4,5 or 6 mm). (Experimental): got generalized unstable periodontitis with a moderately deep pocket (4,5 or 6 mm) will undergo scaling and root surface debritment
  Interventions: Device: Scaling and root surface debritment

INTERVENTIONS:
Device: Scaling and root surface debritment — Patients with 4-6 mm pocket depth were participated in this study; clinical periodontal parameters (BOP, PLI, PPD, CAL) were recorded at the baseline visit. To ensure sampling accuracy, From the site two papers with GCF were sampled. Following sample collecting for GCF, Every patient received comprehensive mouth supragingival scaling with an ultrasonic scaler (WoodpEEKer® UDS-K) along with dental hygiene recommendations. One week later, the sites were irrigated with normal saline after being scaled and root planed (ScRp) with Gracey curette. Following completion of subgingival instrumentation, each patient returned to the clinic following 1 and 3 months for periodontal parameter recording and GCF collection. Throughout these sessions, every patient received reinstruction to engage in self-oral hygiene practices.
  Other Names: Scaling and root planing

SUMMARY:
Periodontitis is a chronic inflammatory disease resulting from bacterial invasion. Endothelin (ET-1) is a potent vasoconstrictor critical in the pathophysiology of periodontal diseases.

Aim The present study aimed to measure the ET-1 concentrations in gingival crevicular fluid (GCF) at baseline, one and three months subsequently to non-surgical periodontal therapy.

Material and methods Designed as a clinical trial, 24 periodontitis individuals will be voluntarily consented to participate. Following non-surgical periodontal treatment, GCF samples will be collected to determine the amount of endothelin-1 at baseline, one, and three months. Clinical periodontal parameters will be recorded.

DETAILED DESCRIPTION:
Periodontitis is a chronic inflammatory disease resulting from bacterial invasion. Endothelin (ET-1) is a potent vasoconstrictor critical in the pathophysiology of periodontal diseases.

Aim The present study aimed to measure the ET-1 concentrations in gingival crevicular fluid (GCF) at baseline, one and three months subsequently to non-surgical periodontal therapy.

Material and methods Designed as a clinical trial, 24 periodontitis individuals will be voluntarily consented to participate. Following non-surgical periodontal treatment, GCF samples will be collected to determine the amount of endothelin-1 at baseline, one, and three months. Clinical periodontal parameters will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* systemically healthy
* Generalized unstable periodontitis with a moderately deep pocket (4,5 or 6 mm)

Exclusion Criteria:

* subjects who wore dental prosthesis
* teeth with grade II mobility,
* alcoholic and smoker, had treated caries
* underwent periodontal therapy within the last four months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
PPD | 3 months recall visits
  changes in PPD after non-surgical periodontal treatment.
CAL | 3 months recall visits
  changes in CAL after non-surgical periodontal treatment.

SECONDARY OUTCOMES:
ET-1 | 3 months recall visits
  change in GCF level of Endothelin-1 in 1- and 3- month following the periodontal treatment

IPD SHARING:
Plan to Share IPD: Undecided